CLINICAL TRIAL: NCT06819306
Title: The Effect of Hedia Diabetes Assistant on TiMe-in-range in People With Type 1 Diabetes and Sub-Optimal Glycemic Control in France - A Randomised Controlled Trial.
Acronym: TEMPO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hedia ApS (Industry)
Collaborators: Kyomed (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-A02199-38
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes Mellitus (T1DM)
Keywords: Bolus calculator; Glycemic control; Digital health
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hedia Diabetes Assistant in addition to standard of care treatment (Experimental)
  Interventions: Device: Hedia Diabetes Assistant
- Standard of care treatment (No Intervention)

INTERVENTIONS:
Device: Hedia Diabetes Assistant — Hedia Diabetes Assistant is an insulin bolus calculator app designed to calculate an insulin bolus dose recommendation for people with type 1 or type 2 diabetes on rapid-acting insulin treatment.
  Arms: Hedia Diabetes Assistant in addition to standard of care treatment

SUMMARY:
The goal of this randomized controlled study is to assess the clinical performance and safety of Hedia Diabetes Assistant in adults with type 1 diabetes and suboptimal glycemic control in France. The main question to answer is:

- Does Hedia Diabetes Assistant improve glycemic control? Researchers will compare Hedia Diabetes Assistant in addition to standard treatment to standard treatment alone to see if Hedia Diabetes Assistant can improve glycemic control.

Subjects will:

* Use Hedia Diabetes Assistant in addition to their standard treatment or only use standard treatment for 6 months.
* Visit the clinic once when they are included into the study and will otherwise be followed remotely.
* Fill out questionnaires when they are included and after 6 months.

DETAILED DESCRIPTION:
This randomized controlled trial will enroll 154 adults with type 1 diabetes who have suboptimal glycemic control and are treated with multiple daily injections (MDI) of insulin using a pen-based basal-bolus regimen. Subjects must be using a continuous glucose monitor (CGM) as part of their standard care and be telemonitored.

The study will be conducted at multiple centres in France, with each subject followed for a total duration of six months. During this period, they will have one in-person visit and two follow-up assessments conducted via phone. Data will be collected through the telemonitoring platform.

Subjects will be randomly assigned to either the intervention or control group. The intervention group will use the Hedia Diabetes Assistant in addition to their standard treatment for six months, while the control group will continue with their standard treatment.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent

* Aged ≥ 18 years at the time of signing the informed consent
* Ability to understand, speak and read French fluently
* Diagnosed with type 1 diabetes > 12 months prior to the day of screening TIR <70% of last 14 days or HbA1c >53 mmol/mol (7%) measured within the last month
* Subject must have the cognitive and physical skills to use mobile applications
* Access to a smartphone with iOS version 16 and up or Android version 12 and up
* Treated with the same pen-based insulin regimen with basal insulin (insulin glargine, degludec, or detemir) and rapid-acting insulin (insulin aspart, lispro, glulisine) for at least the three preceding months
* rtCGM use ≥ 1 month from screening date with ≥70% measurements for the last ≥ 14 days
* Willing to use the same type of CGM for the duration of the clinical investigation
* Willing to be telemonitored during the study period
* If female participants of childbearing potential; willing to have a pregnancy test performed and to use a highly effective method of contraception
* Affiliated to the French social security system

Exclusion Criteria:

* Use of human insulin or premixed insulin
* Using a bolus calculator as a part of standard of care treatment at the time of screening
* If the principal investigator deems that subjects are not healthy, not capable of completing the investigation or in other ways deemed unfit for participation in the investigation
* Ongoing participation in other interventional clinical trials or investigations during the investigation period if the principal investigator deems this to potentially affect the safety, clinical performance and/or any study outcomes
* Female who is pregnant, breast-feeding or intends to be pregnant during the investigation period
* Participant under guardianship, conservatorship, safeguard of justice, or any other legal protection measure for a vulnerable adult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time in range | From 14 days before enrollment to the end of treatment at 26 weeks
  Glucose between 3.9 and 10 mmol/L (70 to 180 mg/dL)

SECONDARY OUTCOMES:
Time above range | From 14 days before enrollment to the end of treatment at 26 weeks
  Glucose > 10.0 mmol/L (> 180 mg/dL)
HbA1c | From enrollment to the end of treatment at 26 weeks
Mean sensor glucose | From 14 days before enrollment to the end of treatment at 26 weeks
Glucose Management Indicator (GMI) | From 14 days before enrollment to the end of treatment at 26 weeks
Coefficient of Variation (CV) | From 14 days before enrollment to the end of treatment at 26 weeks
SD of mean glucose | From 14 days before enrollment to the end of treatment at 26 weeks
Time below range | From 14 days before enrollment to the end of treatment at 26 weeks
  Glucose < 3.9 mmol/L (< 70 mg/dL)
Diabetes Treatment Satisfaction | From enrollment to the end of treatment at 26 weeks
  Diabetes Treatment Satisfaction is measured by the Diabetes Treatment Satisfaction Questionnaire
WHOQoL-BREF | From enrollment to the end of treatment at 26 weeks
  Quality of life is measured by the WHOQoL-BREF questionnaire.

OTHER OUTCOMES:
Time above range level 2 | From 14 days before enrollment to the end of treatment at 26 weeks
  Glucose > 13.9 mmol/L (> 250 mg/dL)
Time in tight range | From 14 days before enrollment to the end of treatment at 26 weeks
  Glucose between 3.9 - 7.8 mmol/L (70-140 mg/dL)
Number of hypoglycemic events | From 14 days before enrollment to the end of treatment at 26 weeks
  Number of episodes with glucose < 3.9 mmol/L (< 70 mg/dL) defined as lasting at least 15 minutes.
Time below range level 2 | From 14 days before enrollment to the end of treatment at 26 weeks
  Glucose < 3.0 mmol/L (< 54 mg/dL)
Number of extended hyperglycemic events | From 14 days before enrollment to the end of treatment at 26 weeks
  Number of episodes with glucose > 13.9 mmol/L (> 250 mg/dL) lasting at least 120 minutes
Number of extended hypoglycemic events | From 14 days before enrollment to the end of treatment at 26 weeks
  Number of epsiodes with glucose < 3.9 mmol/L (< 70 mg/dL) lasting at least 120 minutes.
Proportion with time in range | From 14 days before enrollment to the end of treatment at 26 weeks
  Proportion with glucose between 3.9 - 10.0 mmol/L (70 - 140 mg/dL)
Proportion with ≥5% points improvement in time in range from baseline | From 14 days before enrollment to the end of treatment at 26 weeks
Proportion with ≥10% points improvement in time in range from baseline | From 14 days before enrollment to the end of treatment at 26 weeks
Proportion with time below range < 3.9 mmol/L (< 70 mg/dL) for <4% of the time | From 14 days before enrollment to the end of treatment at 26 weeks
Proportion with time below range < 3.0 mmol/L (< 54 mg/dL) for <1% of the time | From 14 days before enrollment to the end of treatment at 26 weeks
Proportion with time above range >10.0 mmol/L (> 180 mg/dL) for <25% of the time | From 14 days before enrollment to the end of treatment at 26 weeks
Proportion with time above range >13.9 mmol/L (> 250 mg/dL) for <5% of the time | From 14 days before enrollment to the end of treatment at 26 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Hospices Civils de Lyon, Lyon
  - Centre hospitalier universitaire de Nantes, Nantes
  - Centre hospitalier universitaire de Nîmes, Nîmes
  - Hôpital Bichat - Claude-Bernard, Paris
  - Centre hospitalier universitaire de Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: No